CLINICAL TRIAL: NCT03156270
Title: A Prospective, Non-Randomized Study to Evaluate Treatment Outcome of Nasal Airway Obstruction Using the Aerin Medical Vivaer™ Stylus
Brief Title: Treatment Outcome Using Vivaer Stylus to Treat Nasal Airway Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aerin Medical (Industry)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP423
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Results first posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2019-10

CONDITIONS: Nasal Obstruction
Keywords: nasal valve; nasal airway obstruction
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Vivaer Stylus Treatment (Experimental): Thermal treatment of the submucosal tissue including cartilage in the internal nasal valve area
  Interventions: Device: Vivaer Stylus

INTERVENTIONS:
Device: Vivaer Stylus — Stylus used to deliver low-power, temperature-controlled, radiofrequency energy to the tissues of the internal nasal valve area
  Other Names: Aerin Medical Stylus

SUMMARY:
This study evaluates subjective and objective measures of treatment outcome after using the Aerin Medical Vivaer™ Stylus to treat nasal obstruction

DETAILED DESCRIPTION:
This is a non-significant risk, prospective, non-randomized study to evaluate subjective and objective measures of nasal obstruction both before and after treatment with the Vivaer Stylus. The Stylus is used to deliver radiofrequency (RF) energy to the nasal valve area to improve symptoms in those diagnosed with nasal airway obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Complaints of nasal obstruction for at least 1 year
* Failed maximum medical therapy (4-6 weeks of steroids)
* Nasal Obstruction Symptom Evaluation (NOSE) score of ≥ 60 at Baseline
* Nasal valve is a primary or significant contributor to the subject's nasal obstruction as determined by the study investigator (based on clinical presentation, physical examination, nasal endoscopy, etc.) and the subject has a positive response to any of the following temporary measures (based on patient history or during office exam):

  1. Use of external nasal dilator strips (e.g., Breathe Right Strips)
  2. Q-Tip test (manual intranasal lateralization)
  3. Use of nasal stents
  4. Cottle Maneuver (manual lateral retraction of the cheek)

Exclusion Criteria:

* Prior surgical treatment of the nasal valve
* Rhinoplasty, septoplasty, inferior turbinate reduction or other surgical nasal procedures within the past three (3) months
* Severe and/or chronic sinusitis, recurrent sinusitis, or allergies leading to nasal obstruction and currently requiring oral corticosteroid therapy
* Severe case of any of the following: septal deviation, turbinate hypertrophy, polyps, or ptotic nose tip believed to be the primary contributor to the subject's nasal obstruction symptoms and warranting surgical intervention
* Known or suspected allergies or contraindications to the anesthetic agents and/or antibiotic medications to be used during the study procedure session
* Known or suspected to be pregnant, or is lactating
* Other medical conditions which in the opinion of the investigator could predispose the subject to poor wound healing or increased surgical risk

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Otto, MD, Principal Investigator — The Ohio State Eye and Ear Institute
Locations (1):
- The Ohio State Eye and Ear Institute, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with a history of chronic nasal obstruction for at least 1 year were prospectively enrolled at this tertiary academic center.
Period: Overall Study
Arm/Group | Vivaer Stylus Treatment
Started | 20
Completed | 18
Not Completed | 2
Not completed — Failed pre-treatment screening | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Includes all subjects treated with the Vivaer Stylus who were evaluated 90 days post-treatment
Groups:
- Subjects Followed Through 90 Days: Patient cohort includes all subjects treated with the Vivaer Stylus who were evaluated 90 days post-treatment
Arm/Group | Subjects Followed Through 90 Days
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (17.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black or African American | 1
  White | 16
Region of Enrollment [Number; unit: participants]
  United States | 18
Nasal Obstruction Symptom Evaluation (NOSE) score [Mean (Standard Deviation); unit: score on a scale] — The Nasal Obstruction Symptom Evaluation (NOSE) scale is a validated disease-specific health status outcomes instrument, used to assess severity of nasal obstruction symptoms. Score ranges from 0 to 100. Higher scores indicate increased symptoms/symptom severity.
  score on a scale | 78.9 (11.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in NOSE Score
Description: Mean change in Nasal Obstruction Symptom Evaluation (NOSE) score from baseline to 90 days post-study procedure. Improvement (90 day score - baseline score) is signified by a negative value.
  The Nasal Obstruction Symptom Evaluation (NOSE) scale is a validated disease-specific health status outcomes instrument, used to assess severity of nasal obstruction symptoms. Score ranges from 0 to 100. Higher scores indicate increased symptoms/symptom severity.
Time Frame: Baseline, 90 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subjects Followed Through 90 Days
Number analyzed (Participants) | 18
units on a scale | -44.5 (27.0)

2. Primary Outcome: Change in VAS of Nasal Obstruction
Description: Change in visual-analog scale (VAS) of nasal obstruction severity as perceived by the subject from baseline to 90 days post-study procedure. Improvement (90-day score - baseline score) is signified by a negative value.
  The visual-analog scale (VAS) of nasal obstruction is presented to the subject as a 10cm line anchored on each end by verbal descriptors: 0 = No Obstruction and 10 = Completely Obstructed. The subject is asked to place a vertical mark on the line to show the level of nasal obstruction they feel. The distance between 0 and the vertical mark made by the subject is measured and the results is expressed in centimeters. Higher scores indicate more severe obstruction.
Time Frame: Baseline, 90 days
Population: Includes all subjects treated with the Vivaer Stylus who were evaluated 90 days post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subjects Followed Through 90 Days
Number analyzed (Participants) | 18
units on a scale | -2.6 (2.2)

3. Other Pre Specified Outcome: Change in Peak Nasal Inspiratory Flow
Description: Peak inspiratory flow measurements of nasal physical resistance
Time Frame: Baseline, 90 days
Measure: Mean (Standard Deviation); unit: ml/sec
Groups:
- Subjects Followed Through 90 Days - Baseline Data; Subjects Followed Through 90 Days - 90 Day Data: Patient cohort includes all subjects treated with the Vivaer Stylus who were evaluated 90 days post-treatment
Arm/Group | Subjects Followed Through 90 Days - Baseline Data | Subjects Followed Through 90 Days - 90 Day Data
Number analyzed (Participants) | 18 | 18
ml/sec | 60.2 (34.5) | 72.4 (43.7)

ADVERSE EVENTS:
Time Frame: From procedure through 90-day evaluation
Description: Subjects were queried for adverse events after the procedure and at the 90-day evaluation visit. Details of events were documented on a standardized case report form.
Arm/Group | Subjects Followed Through 90 Days
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 6/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Followed Through 90 Days (N=18)
Orthopedic injury or surgery (Musculoskeletal and connective tissue disorders) | 2 (6)
Sinusitis (Infections and infestations) | 2 (3)
Dental treatments (Musculoskeletal and connective tissue disorders) | 2 (3)
Body rash (Infections and infestations) | 1 (1)
Colonoscopy with polyp removal (General disorders) | 1 (1)
Bulb on nostril with diminished airflow (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI/Institution will provide Sponsor with a copy of any proposed manuscripts or other material for publication thirty (30) days prior to publication for review and comment. Sponsor's comments shall be given due consideration by PI/Institution. Publication may be delayed at Sponsor's written request for a period not to exceed sixty (60) days if it contains a disclosure of an invention(s) on which either party desires to file a patent.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT03156270/Prot_SAP_000.pdf